CLINICAL TRIAL: NCT03674242
Title: A Randomized Phase 2/3 Study of Eryaspase in Combination With Gemcitabine and Carboplatin Chemotherapy Versus Chemotherapy Alone for the Treatment of Patients With Metastatic or Locally Recurrent Triple-Negative Breast Cancer
Brief Title: Study of Eryaspase in Combination With Chemotherapy Versus Chemotherapy Alone for the Treatment of TNBC (TRYbeCA-2)
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: sponsor decision
Sponsor: ERYtech Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GRASPA-TNBC-2018-02
Record Dates: First submitted 2018-09-14; First posted 2018-09-17 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — eryaspase; Erythrocyte Count; Gemcitabine; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eryaspase plus Chemotherapy (Experimental): eryaspase 100 U/kg dosed at Day 1 and Day 8 of each 3-week cycle in combination with
  * Gemcitabine IV infusion 1000 mg/m2, Day 1 and Day 8.
  * Carboplatin IV infusion at a calculated area under the curve (AUC) of 2.0 (AUC2), Day 1 and Day 8.
  Interventions: Drug: eryaspase (L-asparaginase encapsulated in red blood cells); Drug: Gemcitabine; Drug: Carboplatin
- Chemotherapy alone (Active Comparator): Gemcitabine plus carboplatin dosed at Day 1 and Day 8 of each 3-week cycle
  Interventions: Drug: Gemcitabine; Drug: Carboplatin

INTERVENTIONS:
Drug: eryaspase (L-asparaginase encapsulated in red blood cells) — IV infusion 100 U/kg
  Other Names: ERY001, GRASPA
  Arms: Eryaspase plus Chemotherapy
Drug: Gemcitabine — IV infusion 1000 mg/m2
  Other Names: Gemzar
Drug: Carboplatin — IV infusion AUC2
  Other Names: Paraplatin

SUMMARY:
This is an open-label, multicenter, randomized, Phase 2/3 study in patients with locally recurrent or metastatic triple-negative breast cancer (TNBC) with no more than one prior systemic therapy for locally recurrent or metastatic disease.

DETAILED DESCRIPTION:
The study will consist of 2 parts:

* Part 1 is an open-label, multicenter, randomized Phase 2 exploratory study that will investigate the clinical activity of the combination of eryaspase and gemcitabine/carboplatin in patients with locally recurrent or metastatic TNBC. Data analysis of Part 1 will inform choices for the final design and patient population in Part 2 (Phase 3 study). Patients recruited into Part 1 will not be included in the Intent-to-Treat patient (ITT) population of Part 2 of the study.
* Part 2 will be a randomized Phase 3 study designed to evaluate the efficacy of the combination of eryaspase and gemcitabine/carboplatin in TNBC patients. The current protocol will focus on Part 1.

Part 1 is the focus of the current protocol, with a primary endpoint of DCR. DCR data as determined by an IRR will determine whether or not proceeding to Part 2 is warranted. If so, Part 2 will be implemented via a major amendment to the protocol. Meanwhile, sites will remain open with the expectation that Part 2 will be activated

After providing informed consent and completing the screening assessments, patients who meet all inclusion and no exclusion criteria will be randomized in a 1:1 ratio to one of the following treatment arms:

* Arm A (experimental arm): eryaspase 100 U/kg on Days 1 and 8 of combination chemotherapy with gemcitabine/carboplatin, or
* Arm B (control arm): gemcitabine/carboplatin combination.

Treatment will continue until objective disease progression, unacceptable toxicity, or the patient's withdrawal of consent.

A survival follow-up period will include the collection of survival, progression of disease if applicable, subsequent anti-cancer therapy every 12 weeks (± 1 week)

ELIGIBILITY:
Inclusion Criteria:

1. Female or male, 18 years of age or older.
2. Histologically or cytologically confirmed diagnosis of invasive breast cancer.
3. Metastatic or locally recurrent inoperable breast cancer with no more than one prior systemic therapy.
4. Diagnosis (original primary tumor or subsequent relapse) of triple negative breast cancer, defined as the absence of expression of the following receptors in the primary and/or metastatic tumor tissue:

   * HER2 protein over-expression and/or gene amplification
   * Estrogen receptor (ER), defined as <1% staining by IHC (2).
   * AND progesterone receptors (PgR), defined as <1% staining by IHC.
5. Measurable lesion(s) per RECIST 1.1.
6. Available archival or fresh tumor tissue.
7. Adequate performance status (PS) score.
8. Life expectancy of >12 weeks according to the Investigator's clinical judgment.
9. Females of childbearing potential must have a negative pregnancy test at screening and an additional pregnancy test prior to first dose. Females of childbearing potential must agree to use a highly effective method of contraception during treatment and for at least 6 months after the last dose of study treatment.
10. Adequate laboratory parameters at baseline (obtained <14 days prior to randomization)
11. Patients must be able to understand and comply with the conditions of the protocol and must have read and understood the consent form and provided written informed consent.

Exclusion Criteria:

1. Pregnant or lactating females.
2. Known BRCA1 or BRCA2 mutation carrier.
3. Bone as the only site of disease.
4. Presence of untreated symptomatic central nervous system (CNS) metastases as determined by MRI or CT scan performed during screening.
5. Prior radiotherapy to the only area of measurable disease.
6. Prophylactic use of supportive bone-modifying therapy for skeletal-related events (e.g., bisphosphonate, pamidronate, or denosumab), unless treatment is initiated prior to or within 7 days after randomization.
7. History of recent clinical pancreatitis, according to revised Atlanta criteria, within 3 months of randomization.
8. Neurosensory neuropathy >Grade 2 at baseline.
9. Known history of infection with human immunodeficiency virus (HIV) and/or active infection with hepatitis B or hepatitis C.
10. Known hypersensitivity to gemcitabine, platinum compounds or asparaginase.
11. Patients who have received live or live attenuated vaccines within 3 weeks of randomization.
12. Pre-existing coagulopathy (e.g. hemophilia).
13. History of other malignancies except: adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, or other solid tumors curatively treated with no evidence of disease for >2 years.
14. Any other severe acute or chronic condition/treatments that may increase the risk of study participation
15. Receiving therapy in a concurrent clinical study. Patients must agree not to participate in any other interventional clinical studies during their participation in this trial while on study treatment. Patients taking part in surveys or observational studies are eligible to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Disease Control Rate (DCR) | 1 year after last patient randomized
  To determine whether the addition of eryaspase to gemcitabine and carboplatin improves the disease control rate (DCR) by modified Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as determined by an independent radiological review (IRR) in patients with locally recurrent or metastatic triple-negative breast cancer (TNBC) compared with chemotherapy alone.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | 1 year after last patient randomized
  To compare the DCR between the two treatment arms as determined by the Investigator's assessment.
Objective response rate (ORR) | 1 year after last patient randomized.
  To compare the objective response rate (ORR) between the two treatment arms as determined by the independent radiological review (IRR).
Progression-Free Survival (PFS) | 1 year after last patient randomized.
  To compare progression-free survival (PFS) between the two treatment arms.
Duration of Response (DoR) | 1 year after last patient randomized.
  To compare the duration of response (DoR) between the two treatment arms.
Overall Survival (OS) | 1 year after last patient randomized.
  To compare overall survival (OS) between the two treatment arms.
Incidence of treatment emergent adverse events as assessed by CTCAE v5.0 | Collected from time of informed consent until 30 days after last study treatment.
  To evaluate the safety and tolerability of eryaspase in combination with chemotherapy versus chemotherapy alone by assessing the number of patients with treatment emergent adverse events per CTCAE v5.0.
Clinical response assessed by F-18 fluorodeoxyglucose positron emission tomography (FDG-PET) imaging | Collected at baseline and within 3 days of the end of Cycle 1 in all patients.
  To evaluate the change in F-18 fluorodeoxyglucose (FDG) tumor uptake as a predictor of clinical response following one cycle of treatment with eryaspase and chemotherapy.
Eryaspase induced immunogenecity | Samples will be collected pre-dose at Cycle 1 Day 1 and pre-dose at Cycle 3 Day 1 (each Cycle is 21 days)
  To determine the anti-asparaginase antibodies titer.
Biomarkers potentials in predicting eryaspase activity. | Tissue samples will be collected at baseline. Blood samples for biomarker analysis will be collected during screening, at Cycle 1 Day 1 and Day 8, and at Day 1 of every second cycle ( each is 21 days) until End of Treatment (EOT) visit.
  To determine DNA, RNA and protein levels present in tumor tissues and blood samples.
Pharmacokinetics of eryaspase | Samples will be collected the first day (D1) and the eight day (D8) of Cycle 1 and Cycle 3 treatment (each Cycle is 21 days) and at End of treatment (EOT)
  To determine total and plasma asparaginase activity (U/L)
Pharmacodynamics of eryaspase | Samples will be collected the first day (D1) and the eight day (D8) of Cycle 1 and Cycle 3 treatment (each Cycle is 21 days) and at End of treatment (EOT)
  To determine plasma concentrations of asparagine and glutamine (µmol/L)

CONTACTS AND LOCATIONS:
Locations (16):
- Belgium (5):
  - ZNA Middelheim, Antwerp
  - Institut Jules Bordet, Brussels
  - UZ Brussel, Brussels
  - Grand Hôpital de Charleroi asbl, Charleroi
  - Clinique Sainte-Elisabeth, Namur
- Hungary (3):
  - Debreceni Egyetem - Klinikai Kozpont - Onkologiai Klinika, Debrecen
  - Bacs Kiskun Megyei Korhaz, Kecskemét
  - Jasz-Nagykun-Szolnok Megyei Hetenyi Geza Korhaz-Rendelointezet, Szolnok
- Spain (8):
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Universitario Germans Trias i Pujol, Badalona
  - Hospital Universitario Arnau Vilanova, Lleida
  - Fundacion Jimenez Diaz, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Quirón Madrid, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Virgen del Rocio, Seville